CLINICAL TRIAL: NCT04631302
Title: Work Engagement and Well-being Study (SWELL): A Randomised Controlled Feasibility Trial Evaluating the Effects of Mindfulness Versus Light Physical Exercise at Work
Brief Title: The Work Engagement and Wellbeing Study
Acronym: SWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020.Vainre_Swell
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Mindfulness; Exercise
Keywords: Mindfulness; physical exercise; wellbeing; workplace; web-based intervention
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blind to participant allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: Be Mindful
- Light Physical Exercise (Active Comparator)
  Interventions: Behavioral: Light exercise course

INTERVENTIONS:
Behavioral: Be Mindful — Be mindful is an online course run by the Mental Health Foundation and Wellmind Media. It was developed together with British mindfulness instructors and offers access to its course materials and instructional videos through a website (http://www.bemindfulonline.com).
  The course consists of 11 sessions led by two mindfulness teachers, one female, one male. Using a variety of media (videos, assignments, audio tracks and e-mails), participants are taught to use formal as well as informal mindfulness techniques. The course lasts 4 weeks. For each week, participants are asked to do a daily formal mediation practice (up to 30 minutes but it varies from week to week) and one or two informal exercises.
  Arms: Mindfulness
Behavioral: Light exercise course — The control condition involves light physical exercises aimed at increasing mobility, reducing stiffness, improving circulation, and avoiding pain or repetitive strain injuries that may result from sedentary or repetitive tasks common in office environments. The exercises will include simple whole-body slightly aerobic exercises such as rotation of limbs and stretching. The course was developed by Dr Julieta Galante, a public health doctor, together with an expert in body posture re-education and body techniques.
  The course is designed to match with the mindfulness intervention condition in duration and media (length of videos, amount of written instructions). It also replicates the encouraged use of short breaks (of seconds or minutes) throughout the workday to focus on wellbeing, as occurs in mindfulness.
  Other Names: Physical exercise
  Arms: Light Physical Exercise

SUMMARY:
Mindfulness and exercise are both widely used to improve mental health and well-being. Some people find that these activities also improve their ability to focus. This study aims to find out whether mindfulness and light exercise could be similarly effective in improving mental wellbeing and engagement at work. The study further investigates the cognitive processes (e.g., memory and attention skills) that might improve as a result of mindfulness and exercise.

DETAILED DESCRIPTION:
Mental illness is a major cause of disability worldwide[1]. Much of the adult population is employed and spends 28% of their waking hours doing paid work[2,3]. The occupational environment is therefore an opportune location for preventative mental health interventions. A growing number of employers provide programmes to improve well-being and work performance.

Mindfulness is typically defined as "the awareness that emerges through paying attention on purpose, in the present moment, and non-judgmentally to the unfolding of experience moment by moment". Practising such awareness has been linked to reduction in symptoms of anxiety, depression, and stress in community populations. There is also evidence that mindfulness could improve life satisfaction, overall well-being, and quality of life.

It has also been argued that mindfulness may yield workplace benefits beyond well-being. Mindfulness has been suggested to improve work performance, reduce the negative effects of multitasking, and enhance self-regulation of thoughts, emotions and behaviours. Empirical evidence to support these suggestions, however, is scarce. Furthermore, the mechanisms through which mindfulness impacts work performance are not clear. Understanding mechanisms of change (a) would help to design better, more targeted interventions, (b) would improve our attempts to assess MBPs via selection of more stringent control interventions and (c) may promote a personalised medicine approach by informing understanding of what works for whom and in which context.

Current literature suggests that MBPs could improve work performance through increased mental well-being and/or cognitive control over emotional material. A definitive randomised controlled trial is needed to evaluate these potential mechanisms. However, methodological uncertainties need clarification to inform the design of such a trial. We aim to conduct a feasibility trial to clarify these uncertainties and complete a preliminary investigation of the relationships between mindfulness training, workplace performance and the proposed mechanisms of action: mental well-being and cognitive control.

This feasibility trial will:

1. Estimate the between-groups effect size for the effect of mindfulness, relative to a light exercise control condition, on our primary outcome of work performance, in order to inform power calculation for a larger trial;
2. Explore whether improved cognitive control and/or enhanced mental health could be potential mechanisms underlying the effect of mindfulness on work performance;
3. Determine procedural feasibility of a later stage trial by evaluating the willingness of the participants to be randomised and other practical implications of running a randomised controlled trial;

ELIGIBILITY:
Inclusion Criteria:

* Employee at one of the participating organisations
* Based in the UK

Exclusion Criteria:

* Is currently on a long-term leave
* Is currently suffering from severe periods of anxiety, depression or hypomania/mania;
* Is experiencing other severe mental illnesses;
* Has had a recent bereavement or major loss;
* Has already completed a mindfulness course or have meditated more than 10 hours in the past 10 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Work Role Functioning Questionnaire (WRFQ). | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  All participants will complete the Work Role Functioning Questionnaire's updated version. It is a 25-item measure to capture the perceived difficulties in meeting work demands. Items are rated on a 5-point scale where 0 is difficult all the time and 5 is difficult none of the time. A 6th option allows participants to denote "does not apply for my job". The subscale and total score are summed, with a minimum score 0 and maximum score 100, with higher scores indicating better work functioning. The questionnaire has not been validated in English but is available in English and validations done in Spain, The Netherlands, Norway, and Brazil have shown good Cronbach alphas (0.7-0.9).
  The primary hypothesis will be evaluated with a time (pre, post) x intervention (mindfulness, light exercise) interaction predicting score on the WRFQ.

SECONDARY OUTCOMES:
Work and Social Adjustment Scale | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Those who said they have experienced health problems will be asked to fill in the Work and Social Adjustment Scale which is widely used in the National Health Service's psychology services in England. It has high internal reliability and sensitivity to treatment effects, comparable to GAD-7 and PHQ-9.
Daily work engagement | Days which participant works during the 4 weeks of intervention. For example, if working full-time and if Monday is Day 1 of intervention then measurements will take place on Day 1...5, Day 8...12, Day 16...20, Day 23...27.
  To get a better understanding of daily fluctuations of work engagement that may occur and whether there are any between-group differences, participants will be asked to complete a short questionnaire about their daily work engagement. The link will be sent to participants' e-mail addresses. We will use a short 5-item version of the Work Role Functioning Questionnaire, which features the following items:
  * Start [work] as soon as you arrived (work scheduling demands)
  * Work without mistakes (Output demands)
  * Repeat the same motions (Physical demands)
  * Concentrate on your work (Mental and social demands)
  * Perform multiple tasks (Flexibility demands) Items are rated on a 5-point scale where 0 is difficult all the time and 5 is difficult none of the time. A 6th option allows participants to denote "does not apply for my job".
Emotional Stop Signal Task: Reaction times (in both, go and stop trials) | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Delivery: Computer-based Stimuli: Images that illustrate negative/neutral social situations are presented. Arrows appear pointing left/right/up.
  Typical trial: At the beginning of each trial, a negative/neural image appears. Afterward, a go-signal appears (left/right arrow) toward which participants need to respond (e.g. press left/right key). On a minority of trials, the go-signal is quickly followed by a stop signal (upwards arrow); these stop-signals follow 20% of go-signals. Participants are required to inhibit their go-response when the stop-signal appears.
Emotional Stop Signal Task: response accuracy (failure or success in inhibiting response) | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Delivery: Computer-based Stimuli: Images that illustrate negative/neutral social situations are presented. Arrows appear pointing left/right/up.
  Typical trial: At the beginning of each trial, a negative/neural image appears. Afterward, a go-signal appears (left/right arrow) toward which participants need to respond (e.g. press left/right key). On a minority of trials, the go-signal is quickly followed by a stop signal (upwards arrow); these stop-signals follow 20% of go-signals. Participants are required to inhibit their go-response when the stop-signal appears.
Emotional Stop Signal Task: variability in reaction time throughout the task (ability to overcome errors). | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Delivery: Computer-based Stimuli: Images that illustrate negative/neutral social situations are presented. Arrows appear pointing left/right/up.
  Typical trial: At the beginning of each trial, a negative/neural image appears. Afterward, a go-signal appears (left/right arrow) toward which participants need to respond (e.g. press left/right key). On a minority of trials, the go-signal is quickly followed by a stop signal (upwards arrow); these stop-signals follow 20% of go-signals. Participants are required to inhibit their go-response when the stop-signal appears.
Probabilistic reverse learning task: learning performance indexed via the proportion of correct responses | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Delivery: Computer-based. Stimuli: Abstract shapes with which participants will have no prior experiences.
  Typical trial: At the beginning of each trial, a negative/neural image from the International Affective Picture System appears. Then, the participants are presented with pairs of stimuli (A-B or C-D). One of the stimuli in the pair is more likely to be rewarded than the other (e.g. selecting A or C is reinforced on 80% of trials). Participants must select one of the stimuli (using key-board presses). Through trial-and-error, participants learn which of the two is correct. Feedback is presented after each response. After a certain number of trials, the contingency of reinforcement changes and another stimulus is reinforced (e.g. B is now reinforced on 80% of trials). This task measure participant's ability to track dynamic changes in their environment and alter their response strategies.
Probabilistic reverse learning task: reaction time | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Delivery: Computer-based. Stimuli: Abstract shapes with which participants will have no prior experiences.
  Typical trial: At the beginning of each trial, a negative/neural image from the International Affective Picture System appears. Then, the participants are presented with pairs of stimuli (A-B or C-D). One of the stimuli in the pair is more likely to be rewarded than the other (e.g. selecting A or C is reinforced on 80% of trials). Participants must select one of the stimuli (using key-board presses). Through trial-and-error, participants learn which of the two is correct. Feedback is presented after each response. After a certain number of trials, the contingency of reinforcement changes and another stimulus is reinforced (e.g. B is now reinforced on 80% of trials). This task measure participant's ability to track dynamic changes in their environment and alter their response strategies.
Probabilistic reverse learning task: accuracy, that is whether the chosen stimulus was the one that was correct. | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Delivery: Computer-based. Stimuli: Abstract shapes with which participants will have no prior experiences.
  Typical trial: At the beginning of each trial, a negative/neural image from the International Affective Picture System appears. Then, the participants are presented with pairs of stimuli (A-B or C-D). One of the stimuli in the pair is more likely to be rewarded than the other (e.g. selecting A or C is reinforced on 80% of trials). Participants must select one of the stimuli (using key-board presses). Through trial-and-error, participants learn which of the two is correct. Feedback is presented after each response. After a certain number of trials, the contingency of reinforcement changes and another stimulus is reinforced (e.g. B is now reinforced on 80% of trials). This task measure participant's ability to track dynamic changes in their environment and alter their response strategies.
Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Subjective well-being will be measured with the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS), a questionnaire designed to capture a broad concept of well-being. In SWEMWBS, each item scored on a five-point scale ranging from 1 (none of the time) to 5 (all of the time). The SWEMWBS internal consistency was α =0.84 in a study in the UK general population (n=27,169).
The Perceived Stress Scale | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  The Perceived Stress Scale (PSS) measures the extent to which the individual has perceived events as uncontrollable and overwhelming in the previous month. Validity and reliability of the PSS have good reports. The PSS consists of 10 items, each answered on a five-point scale ranging from 0 to 4. Higher scores indicate higher stress levels.
Patient Health Questionnaire (PHQ-9) | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  The Patient Health Questionnaire (PHQ-9) is used to assess depression severity during the preceding 2 weeks. The PHQ-9 consists of 9 items answered using a four-point scale, ranging from 0 to 3, and a further item asking about the level of difficulty associated with any checked off items. Scores range from 0 to 27 with cut-off points for depression at 5, 10, 15 and 20 for mild, moderate, moderately severe and severe depression, respectively.
General Anxiety Disorder 7-item Scale (GAD-7) | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  The General Anxiety Disorder 7-item Scale (GAD-7) assesses anxiety during the preceding 2 weeks and has been shown to have good reliability and validity. The items are answered using a four-point scale, ranging from 0 to 3 with total scores ranging from 0 to 21. Higher scores indicate increasing functional impairment with cut-offs at 5, 10 and 15 for mild, moderate and severe anxiety, respectively.
Other health problems | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Single item: "Have you had any health problems in the last 7 days that have affected your ability to work?", with options to pick one or several of the following: physical health problems, mental health problems, other health problems, no problems or prefer not to say. If a participant selects one of the first three options (i.e., they have had problems), they will be asked to briefly describe these problems.
Decentering | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Experiences Questionnaire (EQ) is an 11-item measure of decentering. he items were generated to represent the changes believed to occur as a result of mindfulness practice, including lack of identification with one's thoughts, nonreactivity to negative experiences, and self-compassion. Statements are rated on a 5-point scale (never to all the time). The EQ test scores have an acceptable reliability (alphas .81-.84).
Mindfulness | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Mindful Attention Awareness Scale is a self-report questionnaire consisting of 15 items designed to assess a core characteristic of mindfulness - a receptive state of mind in which attention simply observes what is taking place. Internal consistency is good (α = .82), with good test-retest reliability and convergent validity.

OTHER OUTCOMES:
Retention in the trial | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Number of participants completing measures for each time point
Preferred course | 1 week post-intervention (primary outcome measure);
  Index of which course the participant would have preferred to be randomised to
Engagement in courses | Each of 4 weeks during the intervention.
  To index engagement in courses, we will report the number of people accessing each week's practices.
Regularity in engaging in exercise and mindfulness | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  Self-rated estimate of the amount of time spent on exercise and on mindfulness, separately.
Importance of job to participant | Baseline (pre-intervention); 1 week post-intervention (primary outcome measure); 12-week post-intervention
  1-item self-rated on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Maris Vainre, MA, Principal Investigator — MRC CBU
Locations (1):
- MRC Cognition and Brain Sciences Unit, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Details to be confirmed
Supporting Information: Study Protocol

REFERENCES:
- [Background] Abma F, Bjorner JB, Amick BC 3rd, Bultmann U. Two valid and reliable work role functioning questionnaire short versions were developed: WRFQ 5 and WRFQ 10. J Clin Epidemiol. 2019 Jan;105:101-111. doi: 10.1016/j.jclinepi.2018.09.005. Epub 2018 Sep 22. PMID 30253219
- [Background] Abma FI, van der Klink JJ, Bultmann U. The work role functioning questionnaire 2.0 (Dutch version): examination of its reliability, validity and responsiveness in the general working population. J Occup Rehabil. 2013 Mar;23(1):135-47. doi: 10.1007/s10926-012-9379-8. PMID 22869455
- [Background] Amick BC 3rd, Lerner D, Rogers WH, Rooney T, Katz JN. A review of health-related work outcome measures and their uses, and recommended measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3152-60. doi: 10.1097/00007632-200012150-00010. No abstract available. PMID 11124731
- [Background] Bartlett L, Martin A, Neil AL, Memish K, Otahal P, Kilpatrick M, Sanderson K. A systematic review and meta-analysis of workplace mindfulness training randomized controlled trials. J Occup Health Psychol. 2019 Feb;24(1):108-126. doi: 10.1037/ocp0000146. PMID 30714811
- [Background] Cools R, Clark L, Owen AM, Robbins TW. Defining the neural mechanisms of probabilistic reversal learning using event-related functional magnetic resonance imaging. J Neurosci. 2002 Jun 1;22(11):4563-7. doi: 10.1523/JNEUROSCI.22-11-04563.2002. PMID 12040063
- [Background] Crane RS, Brewer J, Feldman C, Kabat-Zinn J, Santorelli S, Williams JM, Kuyken W. What defines mindfulness-based programs? The warp and the weft. Psychol Med. 2017 Apr;47(6):990-999. doi: 10.1017/S0033291716003317. Epub 2016 Dec 29. PMID 28031068
- [Background] Dane, E. (2011). Paying Attention to Mindfulness and Its Effects on Task Performance in the Workplace. Journal of Management, 37(4), 997-1018. https://doi.org/10.1177/0149206310367948
- [Background] Fresco DM, Moore MT, van Dulmen MH, Segal ZV, Ma SH, Teasdale JD, Williams JM. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. Behav Ther. 2007 Sep;38(3):234-46. doi: 10.1016/j.beth.2006.08.003. Epub 2007 Apr 24. PMID 17697849
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Gallasch CH, Alexandre NM, Amick B 3rd. Cross-cultural adaptation, reliability, and validity of the work role functioning questionnaire to Brazilian Portuguese. J Occup Rehabil. 2007 Dec;17(4):701-11. doi: 10.1007/s10926-007-9103-2. Epub 2007 Oct 2. PMID 17909949
- [Background] Glomb, T. M., Duffy, M. K., Bono, J. E., & Yang, T. (2011). Mindfulness at Work. In A. Joshi, H. Liao, & J. J. Martocchio (Eds.), Research in Personnel and Human Resources Management (Vol. 30, pp. 115-157). Emerald Group Publishing Limited. https://doi.org/10.1108/S0742-7301(2011)0000030005
- [Background] Good, D. J., Lyddy, C. J., Glomb, T. M., Bono, J. E., Brown, K. W., Duffy, M. K., Baer, R. A., Brewer, J. A., & Lazar, S. W. (2016). Contemplating Mindfulness at Work: An Integrative Review. Journal of Management, 42(1), 114-142. https://doi.org/10.1177/0149206315617003
- [Background] Hallingberg B, Turley R, Segrott J, Wight D, Craig P, Moore L, Murphy S, Robling M, Simpson SA, Moore G. Exploratory studies to decide whether and how to proceed with full-scale evaluations of public health interventions: a systematic review of guidance. Pilot Feasibility Stud. 2018 May 28;4:104. doi: 10.1186/s40814-018-0290-8. eCollection 2018. PMID 29854417
- [Background] Health and Safety Executive. (2019). Work-related stress, anxiety or depression statistics in Great Britain, 2019 (Annual Statistics). Health and Safety Executive. https://www.hse.gov.uk/statistics/causdis/stress.pdf
- [Background] Jamieson SD, Tuckey MR. Mindfulness interventions in the workplace: A critique of the current state of the literature. J Occup Health Psychol. 2017 Apr;22(2):180-193. doi: 10.1037/ocp0000048. Epub 2016 Sep 19. PMID 27643606
- [Background] Johansen T, Lund T, Jensen C, Momsen AH, Eftedal M, Oyeflaten I, Braathen TN, Stapelfeldt CM, Amick B, Labriola M. Cross-cultural adaptation of the Work Role Functioning Questionnaire 2.0 to Norwegian and Danish. Work. 2018;59(4):471-478. doi: 10.3233/WOR-182705. PMID 29733048
- [Background] Josefsson, T., Lindwall, M., & Broberg, A. G. (2014). The Effects of a Short-term Mindfulness Based Intervention on Self-reported Mindfulness, Decentering, Executive Attention, Psychological Health, and Coping Style: Examining Unique Mindfulness Effects and Mediators. Mindfulness, 5(1), 18-35. https://doi.org/10.1007/s12671-012-0142-1
- [Background] Kabat-Zinn, J. (2003). Mindfulness-based interventions in context: Past, present, and future. Clinical Psychology: Science and Practice, 10(2), 144-156. https://doi.org/10.1093/clipsy/bpg016
- [Background] Kamerade D, Wang S, Burchell B, Balderson SU, Coutts A. A shorter working week for everyone: How much paid work is needed for mental health and well-being? Soc Sci Med. 2019 Nov;241:112353. doi: 10.1016/j.socscimed.2019.06.006. Epub 2019 Jun 18. PMID 31227212
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Marks, I. M., & Bird, J. (1986). Behavioural psychotherapy: Maudsley pocket book of clinical management (6th ed.). Wright.
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Ramada JM, Serra C, Amick BC 3rd, Abma FI, Castano JR, Pidemunt G, Bultmann U, Delclos GL. Reliability and validity of the work role functioning questionnaire (Spanish version). J Occup Rehabil. 2014 Dec;24(4):640-9. doi: 10.1007/s10926-013-9495-0. PMID 24389721
- [Background] Shapiro, S. L., Astin, J. A., Bishop, S. R., & Cordova, M. (2005). Mindfulness-Based Stress Reduction for Health Care Professionals: Results From a Randomized Trial. International Journal of Stress Management, 12(2), 164-176. https://doi.org/10.1037/1072-5245.12.2.164
- [Background] Shapiro, S. L., Wang, M. C., & Peltason, E. H. (2015). What is mindfulness, and why should organizations care about it? In J. Reb & P. W. B. Atkins (Eds.), Mindfulness in Organizations (pp. 17-41). Cambridge University Press. https://doi.org/10.1017/CBO9781107587793.004
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Zahra D, Qureshi A, Henley W, Taylor R, Quinn C, Pooler J, Hardy G, Newbold A, Byng R. The work and social adjustment scale: reliability, sensitivity and value. Int J Psychiatry Clin Pract. 2014 Jun;18(2):131-8. doi: 10.3109/13651501.2014.894072. Epub 2014 Mar 16. PMID 24527886
- [Derived] Vainre M, Dalgleish T, Watson P, Haag C, Dercon Q, Galante J, Hitchcock C. Work Engagement and Well-being Study (SWELL): a randomised controlled feasibility trial evaluating the effects of mindfulness versus light physical exercise at work. BMJ Ment Health. 2024 Feb 28;27(1):e300885. doi: 10.1136/bmjment-2023-300885. PMID 38423582
- [Derived] Vainre M, Galante J, Watson P, Dalgleish T, Hitchcock C. Protocol for the Work Engagement and Well-being Study (SWELL): a randomised controlled feasibility trial evaluating the effects of mindfulness versus light physical exercise at work. BMJ Open. 2022 Apr 12;12(4):e050951. doi: 10.1136/bmjopen-2021-050951. PMID 35414541